CLINICAL TRIAL: NCT04313764
Title: The Comparison of the Erector Spinae Plane Block and Wound Infiltration on Postoperative Opioid Consumption in Patients Undergoing Laparoscopic Colorectal Surgery
Brief Title: Ultrasound-Guided Erector Spinae Plan Block for Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Medical Doctor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESP Colorectal Surgery
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer; Postoperative Pain
MeSH Terms: conditions — Colorectal Neoplasms; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESPB (Active Comparator): Ultrasound-guided erector spinae plane block with 20 ml %0.25 bupivacaine, per side
  Interventions: Drug: Bupivacaine Hcl 0.25% ESP block
- Group Infiltration (Active Comparator): Wound infiltration with 20 ml %0.25 bupivacaine
  Interventions: Drug: Bupivacaine Hcl 0.25% infiltration

INTERVENTIONS:
Drug: Bupivacaine Hcl 0.25% ESP block — Ultrasound-guided erector spinae plane block with 20 ml %0.25 bupivacaine, per side
  Arms: Group ESPB
Drug: Bupivacaine Hcl 0.25% infiltration — Wound infiltration with 20 ml %0.25 bupivacaine
  Arms: Group Infiltration

SUMMARY:
Colorectal cancer is a common and lethal disease. It still remains the third most common cause of cancer death in women and the second leading cause of death in men. Pain control is an important direction of postoperative management in malignancy surgery. Inadequate pain control increases cardiac and respiratory complications in these critical patients. Erector spinae plane (ESP) block is a recently described regional anesthesia technique that blocks the dorsal and ventral rami of the spinal nerves and the sympathetic nerve fibers. While the ESP block has been shown to provide effective postoperative analgesia after thoracic, and abdominal surgeries.

Our aim in this study was to investigate bilateral thoracic ESP block for providing successful postoperative pain management following colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II-III patients undergoing Colorectal surgery

Exclusion Criteria:

* renal or hepatic insufficiency, chronic pain, patients with an allergic reaction to anesthesia and analgesia drugs to be used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-18 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | Postoperative first 24 hours
  Opioid consumption postroperative period

SECONDARY OUTCOMES:
Visual Analog Pain Score | Postoperative first 24 hours
  Pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Hain E, Maggiori L, Prost A la Denise J, Panis Y. Transversus abdominis plane (TAP) block in laparoscopic colorectal surgery improves postoperative pain management: a meta-analysis. Colorectal Dis. 2018 Apr;20(4):279-287. doi: 10.1111/codi.14037. PMID 29381824
- [Background] Tulgar S, Ahiskalioglu A, De Cassai A, Gurkan Y. Efficacy of bilateral erector spinae plane block in the management of pain: current insights. J Pain Res. 2019 Aug 27;12:2597-2613. doi: 10.2147/JPR.S182128. eCollection 2019. PMID 31695476